CLINICAL TRIAL: NCT02128594
Title: Serosorting Intervention for HIV Negative MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H10-299; R01MH094230 (NIH)
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: STDs
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Standard of Care (Experimental): Standard of care
  Interventions: Behavioral: Serosorting Intervention

INTERVENTIONS:
Behavioral: Serosorting Intervention — Single session, behavioral intervention

SUMMARY:
Men who have sex with men make up a majority of incident HIV infections, however few effective interventions to prevent HIV transmission among this group exist. African American men who have sex with men (AAMSM) are disproportionately infected with STI/HIV and little is understood about how the role of stigma impacts their linkage and retention to health care during treatment. Effective strategies for reducing HIV related risk taking are urgently needed to prevent further spread of the HIV epidemic. The proposed research will test a behavioral intervention, which can be used during routine public health services, designed to reduce HIV risks posed by sexual partner selection strategies. The proposed research will also identify treatment barriers among MSM who test HIV/STI positive. Effective strategies for reducing social barriers to health care treatment rely on a comprehensive and thorough investigation into social barriers that affect AAMSM to effectively engage in medical care. These areas of research will be focused on for the current trial.

DETAILED DESCRIPTION:
Men who have sex with men continue to make up a majority of incident HIV infections. Despite alarmingly high rates of HIV infection, there are few effective interventions to prevent HIV transmission among these men. This five year study, proposed by a New/Early Stage Investigator, consists of a randomized controlled trial to test a behavioral intervention designed to reduce risks for HIV/AIDS posed by sexual partner selection strategies, specifically serosorting, among at-risk HIV negative men who have sex with men in Atlanta, GA. Serosorting - limiting unprotected sexual partners to those of the same HIV status- has emerged as a risk reduction strategy with little input from public health agencies. It is commonly practiced among men who have sex with men to avoid HIV infection. However, engaging in serosorting is a predictor of HIV transmission rather than a reliable form of prevention. Serosorting is ineffective due to several factors, including: multiple flaws in the ability to be certain of own or partner's HIV statuses, the failure of routine HIV tests to detect acute HIV infection, elevated infectiousness due to acute HIV infection, and increased risk for contracting other STIs that can facilitate HIV transmission. We are therefore proposing to test a brief, single-session, Conflict Theory of Decision Making based intervention for use in public health settings. This project uses a novel theory of informed decision making to guide an intervention designed for use in routine services, i.e., HIV post-test counseling. An intervention to address the needs of men who test HIV negative fits well with current efforts to scale up HIV testing, also referred to as seek, test and treat. The proposed research builds on the strengths of a pilot tested, behavioral intervention for addressing serosorting among men who have sex with men. Following screening, informed consent, baseline assessments, and HIV testing (we predict 70 men will test HIV positive), 600 HIV-negative participants will be randomly assigned to receive one of two intervention arms: (a) a serosorting, partner selection intervention, or (b) a time-match, CDC based, post-HIV test counseling, standard-of-care. Participants will be followed over 12-months and assessments will include measures of serosorting beliefs, decisional balance, knowledge of acute HIV infection, HIV status disclosure, and biological (incident STI) and behavioral outcomes (sexual behaviors). This study will test the hypotheses that a brief, single session, serosorting intervention will result in less risk-related serosorting beliefs, greater knowledge/awareness of HIV transmission risk taking, increased HIV status disclosure, reductions in number of sex partners, unprotected sex acts, and incident STIs among intervention participants more so than the control group participants. Moreover, we will test the hypothesis that the intervention will be cost saving when tested in cost-effectiveness analyses. If shown effective, the intervention model will be ready for immediate dissemination to HIV testing services. In a subset of participants, we will test how stigma affects linkage, engagement and retention in care for participants who test HIV/STI positive.

ELIGIBILITY:
Inclusion Criteria:

* Men who have sex with men
* Reside in study area (Atlanta, GA)
* At least 18 years of age
* Other criteria may apply

Exclusion Criteria:

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2012-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Sexually Transmitted Disease | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Eaton, PhD, Principal Investigator — University of Connecticut
Locations (1):
- SHARE Project, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Eaton LA, Kalichman SC, Kalichman MO, Driffin DD, Baldwin R, Zohren L, Conway-Washington C. Randomised controlled trial of a sexual risk reduction intervention for STI prevention among men who have sex with men in the USA. Sex Transm Infect. 2018 Feb;94(1):40-45. doi: 10.1136/sextrans-2016-052835. Epub 2017 Apr 12. PMID 28404766